CLINICAL TRIAL: NCT04164511
Title: Impact of Ice Cream Consumption on Postoperative Rrecovery After Tonsillectomy
Brief Title: Does Ice Cream Help With Post-tonsillectomy Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital Sestre Milosrdnice
Other Study IDs: EP-SLA01
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Tonsillitis; Postoperative Pain; Cryotherapy Effect
Keywords: pediatric; tonsillectomy; ice cream; cryotherapy; postoperative pain
MeSH Terms: conditions — Tonsillitis; Pain, Postoperative | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with post-tonsillectomy ice cream: Pediatric patients undergoing tonsillectomy and receiving 2 daily ice creams for 2 weeks after surgery. Standard analgesic therapy available.
  Interventions: Dietary Supplement: 2 daily standard doses of vanilla-chocolate ice cream (cryotherapy)
- Patients without post-tonsillectomy ice cream: Pediatric patients undergoing tonsillectomy, not receiving any ice cream for 2 weeks after surgery. Standard analgesic therapy available.
  Interventions: Dietary Supplement: 2 daily standard doses of vanilla-chocolate ice cream (cryotherapy)

INTERVENTIONS:
Dietary Supplement: 2 daily standard doses of vanilla-chocolate ice cream (cryotherapy) — The patients will receive 2 daily standard doses of vanilla-chocolate ice cream (cryotherapy) for 2 weeks post-op, with amount of analgesic consumption and subjective pain levels recorded on a VAS scale.

SUMMARY:
Tonsillectomy is one of the most performed procedures in childhood, which carries with it certain postoperative problems, such as the pain of the operated area. Sickness greatly impairs the quality of life in the postoperative period and further reduces food and fluid intake in children, which in turn causes prolonged recovery after surgery. The impact of cooling oropharynx in the form of ice cream consumption as a form of cryotherapy could help reduce the pain, reduce the use of oral analgesic therapy and help in faster recovery after surgery.

Research goal:

The aim of the study is to determine whether the consumption of ice cream, as a form of cryotherapy, influences the rate of postoperative recovery after tonsillectomy and the consumption of oral analgesics in children.

The study was designed as a prospective, randomized, parallel-group, unmasked, and longitudinal study enroling 100 children undergoing tonsillectomy in a tertiary referral center. Of those children, 60 will consume the same ice cream (a combination of vanilla and chocolate as universally acceptable flavors) twice daily, morning and evening, for two weeks after surgery. 40 children will not consume ice cream during the stated period. Parents will be given a questionnaire with a validated VAS Wong-Baker FACES scale (Visual - Analogue - Scale) used by the Zagreb Pediatric Disease Clinic to be completed at home based on communication with the child and containing information on a visual-analogue subjective pain experience in children every morning after eating ice cream and the amount of analgesics the children received during the first two weeks after surgery. There will also be a record of the days when children began to consume food and drink in the same range and quality as before surgery.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most performed procedures in childhood, which carries with it certain postoperative problems, such as the pain of the operated area. Sickness greatly impairs the quality of life in the postoperative period and further reduces food and fluid intake in children, which in turn causes prolonged recovery after surgery. The impact of cooling oropharynx in the form of ice cream consumption as a form of cryotherapy could help reduce the pain, reduce the use of oral analgesic therapy and help in faster recovery after surgery. Also, this research represents the first recorded attempt in the literature to test the myth of the association between tonsillectomy and ice cream in children in a prospective nonrandomized study with parallel intervention groups.

Research goal:

The aim of the study is to determine whether the consumption of ice cream, as a form of cryotherapy, influences the rate of postoperative recovery after tonsillectomy and the consumption of oral analgesics in children.

Research participants:

100 children undergoing tonsillectomy at the Clinic for Otorhinolaryngology and Head and Neck Surgery at the Clinical Hospital Center "Sisters of Mercy" The study was designed as a prospective, randomized, parallel-group, unmasked, and longitudinal study enrolling 100 children undergoing tonsillectomy. Of those children, 60 will consume the same ice cream (a combination of vanilla and chocolate as universally acceptable flavors) twice daily, morning and evening, for two weeks after surgery. 40 children will not consume ice cream during the stated period. Parents will be given a questionnaire with a validated VAS Wong-Baker FACES scale (Visual - Analogue - Scale) used by the Zagreb Pediatric Disease Clinic to be completed at home based on communication with the child and containing information on a visual-analogue subjective pain experience in children every morning after eating ice cream and the amount of analgesics the children received during the first two weeks after surgery. There will also be a record of the days when children began to consume food and drink in the same range and quality as before surgery.

The study will be conducted on children who have tonsillectomy at the Clinic for Otorhinolaryngology and Head and Neck Surgery in the period 12/1/2019 - 6/30/2020, and will include a total of 100 children. Parents will also participate in the research and data collection, in addition to the Clinic doctors involved in this research.

A random coin toss (binary coin-toss method) will determine which child enters the group of children who consume ice cream and which does not.

Data will be collected prospectively at each regular check-up after surgery. The data sought is a subjective feeling of pain, consumption of analgesics in milligrams depending on the type of analgesics, and the postoperative day when the diet returned to normal, preoperative conditions.

There are no risks of participating in the research.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients able to consume ice cream
* sufficient age and dietary status), undergoing tonsillectomy
* informed consent from parents

Exclusion Criteria:

* failure to record data
* incomplete follow-up
* invalid informed consent

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing tonsillectomy in a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Level of post-tonsillectomy pain within first 2 postoperative weeks: VAS scale | 14 days
  Level of post-tonsillectomy pain within first 2 postoperative weeks assessed by VAS scale

SECONDARY OUTCOMES:
Amount of post-tonsillectomy analgesics consumed within first 2 postoperative weeks | 14 days
  Amount of post-tonsillectomy analgesics consumed within first 2 postoperative weeks recorded daily by type and amount (gram or miligram total)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Geber, MD, PhD, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No